CLINICAL TRIAL: NCT06534528
Title: An Open Clinical Study Exploring the Safety, Tolerability, and Preliminary Efficacy of Human Umbilical Cord Mesenchymal Stem Cell Injection in the Treatment of Interstitial Lung Disease (ILD)
Brief Title: Human Umbilical Cord Mesenchymal Stem Cell Injection for the Treatment of Interstitial Lung Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Life Science & Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHLF-MSC-ILD-101
Record Dates: First submitted 2024-07-12; First posted 2024-08-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial Lung Disease; ILD
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Dose1 Group：6.0×10^6 cells/person, single-dose Dose2 Group：3.0×10^7 cells/person, single-dose Dose3 Group：6.0×10^7 cells/person, single-dose Dose4 Group：9.0×10^7 cells/person, single-dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation (Experimental): Four different doses were set, and three subjects in each dose plan received human umbilical cord mesenchymal stem cell injection successively. Each subject received a single dose of 6.0*10^6, 3.0*10^7,6.0*10^7, and 9.0*10^7 cells / person.
  Interventions: Drug: Human umbilical cord mesenchymal stem cell injection

INTERVENTIONS:
Drug: Human umbilical cord mesenchymal stem cell injection — Different doses of human umbilical cord mesenchymal stem cell injection were infused to the focus of patients with idiopathic pulmonary fibrosis through bronchoscope, and the tolerance of subjects to different doses of human umbilical cord mesenchymal stem cell injection was observed, and the curative effect was preliminarily observed.

SUMMARY:
Main objective: To explore the safety and tolerability of human umbilical cord mesenchymal stem cell injection in the treatment of interstitial lung disease (ILD); Secondary objective: To explore the preliminary effectiveness of human umbilical cord mesenchymal stem cell therapy for interstitial lung disease (ILD) and recommend appropriate cell therapy doses for subsequent clinical studies; Exploring the immunogenicity of human umbilical cord mesenchymal stem cell injection in the treatment of interstitial lung disease (ILD).

ELIGIBILITY:
Inclusion Criteria:

* Gender not limited, age ≥ 18 years old (including threshold);
* Clinical diagnosis of interstitial lung disease;
* Blood biochemistry tests must meet the following criteria: alanine aminotransferase (ALT) ≤ 2.5 × ULN, aspartate aminotransferase (AST) ≤ 2.5 × ULN, total bilirubin (TBIL) ≤ 2 × ULN, direct bilirubin (DBIL) ≤ 1.5 × ULN, or creatinine (Cr) ≤ 3 × ULN;
* The diffusion capacity of carbon monoxide (DLCO) (corrected by Hb) in lung function tests within the previous 3 months is 30% to 80% of the expected value (including 30% and 80%); Forced vital capacity (FVC) is 40% to 70% of the estimated value (including 40% and 70%)

Exclusion Criteria:

* Within the first 3 days of enrollment, use high-dose corticosteroids (equivalent to methylprednisolone>240 mg/day) or irregularly use systemic corticosteroids;
* For patients receiving immunosuppressive therapy, unstable background treatment with cyclophosphamide, mycophenolate mofetil/sodium, methotrexate, or other immunosuppressive monotherapy is not allowed (combination therapy is not allowed)
* Diagnose IPF patients who have previously taken drugs that may cause or worsen pulmonary fibrosis;
* Individuals with a history of mechanical ventilation or concurrent infectious pneumonia or asthma within the previous month prior to screening; Patients with airway obstruction disease (FEV1/FVC<0.7 before using bronchodilators); Patients with other clinically significant serious abnormalities in the lungs; Currently requiring oxygen therapy treatment (oxygen therapy time>15h/d);
* Pregnant and lactating women
* Screening for malignant tumors that have occurred within the past 5 years, excluding cervical carcinoma in situ, squamous cell carcinoma of the skin, or basal cell carcinoma that have been previously treated for curative purposes;
* Individuals who have been hospitalized for 3 or more times due to acute exacerbation of ILD or other respiratory diseases within the past year prior to screening
* There is evidence that subjects currently have digestive system, urinary system, cardio cerebrovascular, blood system, nervous system, mental and metabolic diseases that may affect safety, such as type 2 diabetes with poor blood sugar control, hypertension with poor blood pressure control, etc
* have a history of abuse or drug use of psychotropic substances
* individuals allergic to human serum albumin, anesthetics, or their components
* Select participants who have participated in any other clinical trials within the previous 3 months;
* individuals who have previously received stem cell therapy
* Researchers have determined that the expected survival period may be less than 1 year;
* Subjects who cannot tolerate bronchoscopy examination (including but not limited to: active massive hemoptysis; severe hypertension and arrhythmia;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose per dose (MTD) | From the first administration to 4 weeks after administration
  The maximum tolerable dose (MTD) of a single administration depends on whether dose limiting toxicity (DLT) occurs within 4 weeks after the first administration, for example (1) Hematological toxicity of grade 3 and above caused by the treatment of human umbilical cord mesenchymal stem cell injection. There are grade 3 and above non hematological toxic reactions caused by the treatment of human umbilical cord mesenchymal stem cell injection, except for the following cases, (3) Any other toxicity related to cell therapy that is higher than the baseline level is judged as clinically significant and / or unacceptable by the investigator and the sponsor, (4) There are acute exacerbations and serious adverse events (SAE) of IPF related to the treatment of human umbilical cord mesenchymal stem cell injection (which may be related, likely to be related and definitely related)

SECONDARY OUTCOMES:
Preliminary efficacy evaluation：lung function | The 4th, 12th, 24th week after administration
  Changes from baseline in lung function (forced vital capacity, diffusion capacity for carbon monoxide) in the treatment of Interstitial lung disease(ILD), and to recommend the appropriate dose of cell therapy for subsequent clinical studies.
  Forced vital capacity(FVC) in litre(L); Diffusion capacity for carbon monoxide(DLCO) in ml/min/mmHg
Preliminary efficacy evaluation: St. George's respiratory questionnaire(SGRQ) | The 4th, 12th, 24th week after administration
  Changes from baseline in score of St. George's respiratory questionnaire(SGRQ). To study the value of St George s respiratory questionnaire(SGRQ) in evaluating the life quality of patients with ILD, and to recommend the appropriate dose of cell therapy for subsequent clinical studies.
  St. George's respiratory questionnaire(SGRQ) score: Range 0-100,The higher the score, the more severe the impact of the disease on symptoms, activities, and daily life.
Preliminary efficacy evaluation: dyspnea score | The 4th, 12th, 24th week after administration
  Changes from baseline in value of dyspnea score. To study the value of dyspnea score(modified Medical Research Council, mMRC) in evaluating the life quality of patients with ILD, and to recommend the appropriate dose of cell therapy for subsequent clinical studies.
  Dyspnea score(mMRC)：Range 0-4,mMRC levels 0-1 indicate few symptoms, mMRC levels 2-3 indicate multiple symptoms, and level 4 indicates difficulty breathing at the slightest level of activity.
Preliminary efficacy evaluation: cough score | The 4th, 12th, 24th week after administration
  Changes from baseline in value of cough score. To study the value of cough score(Cough Evaluation Test, CET) in evaluating the life quality of patients with ILD, and to recommend the appropriate dose of cell therapy for subsequent clinical studies.
  Cough score(Cough Evaluation Test, CET)：Range 5-25, the higher the score, the more severe the daytime cough, the greater the impact of nighttime cough on sleep, and the greater the impact of cough on daily life and psychology.
Preliminary efficacy evaluation: 6-minute walk test | The 4th, 12th, 24th week after administration
  Changes from baseline in result of 6-minute walk test (grade and distance) in the treatment of Interstitial lung disease(ILD), and to recommend the appropriate dose of cell therapy for subsequent clinical studies.
  Draw a straight distance of 30.5 meters (100 feet) on a flat surface, and place a chair at each end as a marker. The subjects walked back and forth between them, with the pace determined by their own physical abilities. The personnel monitoring on the side report the time every 2 minutes and record any discomfort such as shortness of breath or chest pain that the subject may experience.
Preliminary efficacy evaluation: Frequency of acute exacerbation events | The 4th, 12th, 24th week after administration
  Changes from baseline in Frequency of acute exacerbation events in the treatment of Interstitial lung disease(ILD), and to recommend the appropriate dose of cell therapy for subsequent clinical studies
Preliminary efficacy evaluation: High Resolution Computed Tomography scores(HRCT score) | The 4th, 12th, 24th week after administration
  Changes from baseline in chest High Resolution Computed Tomography scores(Warrick score) in the treatment of Interstitial lung disease(ILD), and to recommend the appropriate dose of cell therapy for subsequent clinical studies.
  HRCT score(Warrick score): Range 0-30,the higher the score, the more severe the lesion type and the wider the lesion range.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]：Blood pressure | The 4th, 12th, 24th week after administration
  Blood pressure in millimeter of mercury(mmHg)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]：Pulse | The 4th, 12th, 24th week after administration
  Pulse in beats per minute
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]：respiration rate | The 4th, 12th, 24th week after administration
  Respiration rate in times/minute
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]：body temperature | The 4th, 12th, 24th week after administration
  Body temperature in centigrade(℃)
Blood routine | The 4th, 12th, 24th week after administration
  White blood cell count (WBC) in 10^9/L; Neutrophil count (Neu) in 10^9/L; Lymphocyte count (Lym) in 10^9/L; Monocyte count (Mon) in 10^9/L; Eosinophil count (Eos) in 10^9/L; Basophil count(Bas) in 10^9/L; Red blood cell count (RBC) in 10^9/L; Platelets(PLT) in 10^9/L; Hemoglobin (HGB) in g/L; Mean corpuscular hemoglobin concentration (MCHC) in g/L; Hematocrit (HCT) in percentage(%); Mean corpuscular volume (MCV) in femtoliter(fL).
Blood biochemistry | The 4th, 12th, 24th week after administration
  Total protein (TP) in g/L; Albumin (ALB) in g/L; Total bilirubin (TBIL) in umol/L, Direct bilirubin (DBIL) in umol/L, Total bile acid (TBA) in umol/L, Creatinine (Cr) in umol/L, Uric acid (UriC) in umol/L; Alanine aminotransferase (ALT) in U/L Aspartate aminotransferase (AST) in U/L; Alkaline phosphatase (ALP) in U/L; Gamma glutamyl transpeptidase (GGT) in U/L; Lactate dehydrogenase (LDH) in U/L; Fasting blood glucose (Glu) in mmol/L; Potassium ions (K+) in mmol/L; Sodium ions (Na+) in mmol/L; Chloride ions (Cl -) in mmol/L; Calcium ions (Ca2+) in mmol/L; Glycated hemoglobin (HbA1c) in percentage(%);
Blood gas analysis | The 4th, 12th, 24th week after administration
  PH; Arterial partial pressure of oxygen (PaO2) in mmHg Arterial partial pressure of carbon dioxide (PaCO2) in mmHg
Concentration of Lung tumor markers | The 4th, 12th, 24th week after administration
  Cytokeratin 19 fragment (CYFRA21-1) in ng/mL; Neuron specific enolase (NSE) in ng/mL; Squamous cell carcinoma antigen (SCC) in ng/mL; Carcinoembryonic antigen (CEA) in ng/mL; Carbohydrate antigen(CA125) in Unit/mL.
Electrocardiogram | The 4th, 12th, 24th week after administration
  Heart rate in beats/minute; PR interval in millisecond(ms) QRS interval in millisecond(ms) QT interval (uncorrected) in millisecond(ms)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maher TM. Interstitial Lung Disease: A Review. JAMA. 2024 May 21;331(19):1655-1665. doi: 10.1001/jama.2024.3669. PMID 38648021
- [Background] Rosas IO, Dellaripa PF, Lederer DJ, Khanna D, Young LR, Martinez FJ. Interstitial lung disease: NHLBI Workshop on the Primary Prevention of Chronic Lung Diseases. Ann Am Thorac Soc. 2014 Apr;11 Suppl 3(Suppl 3):S169-77. doi: 10.1513/AnnalsATS.201312-429LD. PMID 24754826
- [Background] Gille T, Laveneziana P. Cardiopulmonary exercise testing in interstitial lung diseases and the value of ventilatory efficiency. Eur Respir Rev. 2021 Nov 30;30(162):200355. doi: 10.1183/16000617.0355-2020. Print 2021 Dec 31. PMID 34853093
- [Background] Hass R, Kasper C, Bohm S, Jacobs R. Different populations and sources of human mesenchymal stem cells (MSC): A comparison of adult and neonatal tissue-derived MSC. Cell Commun Signal. 2011 May 14;9:12. doi: 10.1186/1478-811X-9-12. PMID 21569606
- [Background] Moodley Y, Atienza D, Manuelpillai U, Samuel CS, Tchongue J, Ilancheran S, Boyd R, Trounson A. Human umbilical cord mesenchymal stem cells reduce fibrosis of bleomycin-induced lung injury. Am J Pathol. 2009 Jul;175(1):303-13. doi: 10.2353/ajpath.2009.080629. Epub 2009 Jun 4. PMID 19497992
- [Background] Averyanov A, Koroleva I, Konoplyannikov M, Revkova V, Lesnyak V, Kalsin V, Danilevskaya O, Nikitin A, Sotnikova A, Kotova S, Baklaushev V. First-in-human high-cumulative-dose stem cell therapy in idiopathic pulmonary fibrosis with rapid lung function decline. Stem Cells Transl Med. 2020 Jan;9(1):6-16. doi: 10.1002/sctm.19-0037. Epub 2019 Oct 15. PMID 31613055
- [Background] Chambers DC, Enever D, Ilic N, Sparks L, Whitelaw K, Ayres J, Yerkovich ST, Khalil D, Atkinson KM, Hopkins PM. A phase 1b study of placenta-derived mesenchymal stromal cells in patients with idiopathic pulmonary fibrosis. Respirology. 2014 Oct;19(7):1013-8. doi: 10.1111/resp.12343. Epub 2014 Jul 9. PMID 25039426
- [Background] Glassberg MK, Minkiewicz J, Toonkel RL, Simonet ES, Rubio GA, DiFede D, Shafazand S, Khan A, Pujol MV, LaRussa VF, Lancaster LH, Rosen GD, Fishman J, Mageto YN, Mendizabal A, Hare JM. Allogeneic Human Mesenchymal Stem Cells in Patients With Idiopathic Pulmonary Fibrosis via Intravenous Delivery (AETHER): A Phase I Safety Clinical Trial. Chest. 2017 May;151(5):971-981. doi: 10.1016/j.chest.2016.10.061. Epub 2016 Nov 24. PMID 27890713